CLINICAL TRIAL: NCT05297474
Title: Structural and Functional Impairment of Multiple Organs in Patients With Systemic Sclerosis: A MR Imaging Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xihai Zhao, Professor, Tsinghua University
Other Study IDs: 12040740374
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Systemic Sclerosis; Multisystem Disorder
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ForIL-2/6/9、5Ht and PON-1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SSc patiant: We recruited 95 patients with systemic sclerosis
  Interventions: Other: MRI
- health control: We recruited 95 healthy people for control
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — No intervention was performed in this study.

SUMMARY:
This study intends to carry out a prospective, multi-center cohort study based on MRI to explore the incidence of structural and functional damage of central, brain and kidney in patiant with SSc and its clinical relevance, and to search for the characteristics of serological markers of structural and functional damage of heart, brain and kidney.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a autoimmune disease of unknown etiology with an estimated global incidence of 0.1‰. SSc characterized by abnormal immune activation, neovascularization, vascular remodeling in pathology, and eventually leads to fibrosis of tissues, skin, and organs [2]. In addition to skin sclerosis, SSc often involved multiple organ involvement, such as finger ulcer, gastroesophageal reflux, interstitial lung disease, pulmonary hypertension, cardiomyopathy, kidney damage, etc. Neuropsychiatric manifestations such as anxiety and depression may also occur in SSc patients. A long-term follow-up study indicated that cardiomyopathy (14%), cardiovascular disease (12%), and kidney injury (4%) were important causes of death in SSc patients. Therefore, early diagnosis and early intervention for multi-organ complications of SSc can significantly prolong the survival time of SSc patients.Magnetic resonance imaging (MRI) is a non-invasive, radiation-free imaging examination method with excellent soft tissue contrast, which can achieve one-stop multi-parameter imaging. At present, MRI has been widely used to accurately diagnose and evaluate the structure and function of organs such as heart, brain and kidney. Previous literature has shown that cardiac MRI can identify cardiac injury in patients with SSc earlier than echocardiography even in the early stage. Meanwhile it can find the abnormalities before clinical symptoms. Therefore, MRI is an effective noninvasive imaging method to evaluate the structural and functional damage of heart, brain and kidney in SSc patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of systemic sclerosis

Exclusion Criteria:

Complicated with other immune disease Claustrophobia Contraindications for MR examination Heart or respiratory failure Diseases that affect MR findings (e.g. rapid atrial fibrillation) Complicated with heart, brain and kidney diseases not caused by SSc（such as diabetic nephropathy and congenital heart disease） Pregnant Disturbance of consciousness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we plan to recruit patients with systemic sclerosis and to explore the incidence and clinical correlation of structural and functional damage of heart, brain and kidney by MRI.The patients will be recruited in China.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of structural and functional disorders of heart, brain and kidney in SSc patients. | 1year.
  The incidence of structural and functional disorders of heart, brain and kidney in SSc patients.

CONTACTS AND LOCATIONS:
Overall Officials: Huilin He, MD, Principal Investigator — Peking Union Medical College Hospital; Chenlin Du, PhD, Principal Investigator — Tsinghua University
Locations (2):
- China (2):
  - Huilin He, Beijing
  - China Center for Biomedical Imaging Research, Department of Biomedical Engineering, Tsinghua University, Beijing

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05297474/Prot_ICF_000.pdf